CLINICAL TRIAL: NCT02064803
Title: Randomized Clinical Trial Comparing Gastric Partitioning Plus Gastro-entero Anastomosis Versus Gastro-entero Anastomosis Only in Patients With Unresectable and Obstructive Distal Gastric Cancer.
Brief Title: Gastric Partitioning Procedure for the Treatment of Unresectable and Obstructive Distal Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP382/13
Record Dates: First submitted 2014-01-31; First posted 2014-02-17 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group: A (Active Comparator): Gastro-entero anastomosis only
  Interventions: Procedure: Gastro-entero anastomosis only
- Experimental: B (Experimental): Gastric partitioning Plus Gastro-entero anastomosis
  Interventions: Procedure: Gastric partitioning Plus Gastro-entero anastomosis

INTERVENTIONS:
Procedure: Gastro-entero anastomosis only — Gastro-entero anastomosis only
  Arms: Control group: A
Procedure: Gastric partitioning Plus Gastro-entero anastomosis — Gastric partitioning Plus Gastro-entero anastomosis
  Arms: Experimental: B

SUMMARY:
The incidence of unresectable and obstructive gastric cancer patients ranges in the literature from 5 to 30 % . In such cases, gastro-entero anastomosis is traditionally performed and can improve the quality of life by relieving the symptoms of impaired oral intake without having a high surgical risk. Unfortunately, up to 25% of these patients may develop impaired gastric emptying syndrome. Gastric partitioning was originally described by Devine in 1925 as a method of antral exclusion and complete division of the stomach accompanied by a gastro-entero anastomosis in the proximal gastric pouch for the management of difficult duodenal ulcers. This procedure has been modified along the years and was adopted for the palliative treatment of gastric cancer. The advantages of the partitioning includes: better gastric emptying, avoidance of direct tumor invasion of the gastro-entero anastomosis, less contact between the ingested food and the tumor with less blood lost and improved survival. Retrospective not randomized studies have been published demonstrating the effectiveness of the procedure.

DETAILED DESCRIPTION:
The first group (Group A) will be considered the control group in which patients will undergo gastro-entero anastomosis. The anastomosis will be pre-colic, along the posterior wall of the stomach with the length of at least 5 cm. The first jejunal loop approximately 40 cm from the angle of Treitz will be used. The anastomosis can be performed manually or with staplers.

The second group (group B) will be considered the intervention group in which patients will undergo gastric partitioning plus gastro-entero anastomosis. The gastric partitioning is done 5 cm proximal to the lesion along the greater curvature towards the lesser curvature above the incisura using linear cutting stapler. The partitioning is performed horizontally and preserve a narrow tunnel along the lesser curvature that is calibrated with a orogastric tube gauge 32. Subsequently, a pre-colic gastro-entero anastomosis is performed in the proximal gastric chamber created by the partitioning. The anastomosis is done along the posterior wall, with at least 5 cm of length using the first jejunal loop approximately 40 cm from the angle of Treitz. The anastomosis can be performed manually or with staplers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal obstructive gastric tumors without indication of curative or palliative resection.
* Obstruction is defined as GOOSS (Gastric outlet obstruction score system) of 2 or less, associated with early vomiting and bloating if the patient try to keep the usual volume of food intake.
* Confirmation that obstruction is gastroduodenal by imaging and Upper Digestive Endoscopy ( EDA )
* Absence of other points of obstruction distal to the gastric tumor
* Histological diagnosis of cancer confirmed by biopsy
* Patients who has signed the informed consent form

Exclusion Criteria:

* Refusal to sign the informed consent form
* Tumors with indication of curative or palliative resection
* Proximal gastric tumors located above the incisura along the lesser curvature
* Tumors that invade the greater curvature above the middle third of the stomach
* Patients with low clinical performance - ECOG (Eastern Cooperative Oncology Group) 3 and 4.
* Obstruction located in the small intestine or colon
* Diffuse peritoneal carcinomatosis with peritoneal carcinomatosis index greater than 12

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline Gastric Outlet Obstruction Score System - GOOSS | 6 months
  Gastric Obstruction measured by the gastric outlet obstruction scoring system (GOOSS). From baseline, participants will be followed every 2 months for the duration of survival, an expected average of less than 6 months

SECONDARY OUTCOMES:
Overall survival | 6 months
  From baseline, participants will be followed every 2 months for the duration of survival, an expected average of less than 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcus K. Ramos, MD, Principal Investigator — Instituto do Câncer do Estado de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil